CLINICAL TRIAL: NCT02734602
Title: Imaging SV2A in Mood Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Irina Esterlis, Assistant Professor, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1511016789
Record Dates: First submitted 2016-03-17; First posted 2016-04-12 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder; Post-Traumatic Stress Disorder
Keywords: depression; post-traumatic stress disorder; sv2a; ketamine; PET
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Depression | interventions — Ketamine; TP63 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single PET scan (No Intervention): Subjects will participate in 1 PET scan (up to 2 if cancelations occur) on the High Resolution Research Tomograph (HRRT), the highest resolution human brain scanner available, or the HR+ will be used to image subjects. Vital signs (blood pressure and pulse) will be obtained before and after radiotracer administration. Venous catheter(s) will be used for IV administration of the radiotracer and for venous blood sampling. An arterial catheter will be inserted by an experienced physician before the PET scan.
- PET scans and ketamine administration (Active Comparator): Subjects will participate in 2-3 PET scans (up to 4 if cancelations occur) on the High Resolution Research Tomograph (HRRT), the highest resolution human brain scanner available, or the HR+ will be used to image subjects. Vital signs (blood pressure and pulse) will be obtained before and after radiotracer administration. Venous catheter(s) will be used for IV administration of the radiotracer and for venous blood sampling. An arterial catheter will be inserted by an experienced physician before the PET scan. After a baseline scan, subjects will be administered a low dose of ketamine for the second scan.
  Bipolar subjects will not participate in any ketamine arms.
  Interventions: Drug: Ketamine
- PET scans for subjects undergoing ketamine treatment (No Intervention): For subjects currently undergoing treatment with ketamine. Subjects will participate in 1-3 PET scans (up to 4 if cancelations occur) on the High Resolution Research Tomograph (HRRT), the highest resolution human brain scanner available, or the HR+ will be used to image subjects. Vital signs (blood pressure and pulse) will be obtained before and after radiotracer administration. Venous catheter(s) will be used for IV administration of the radiotracer and for venous blood sampling. An arterial catheter will be inserted by an experienced physician before the PET scan. Baseline scan will occur prior to initiation of ketamine treatment. Subsequent scans will occur after several treatments with ketamine and after completion of treatment.
  Bipolar subjects will not participate in any ketamine arms.

INTERVENTIONS:
Drug: Ketamine — Ketamine will be administered after the initial PET scan for subjects participating in the ketamine aim.
  Other Names: Ket
  Arms: PET scans and ketamine administration

SUMMARY:
This study is designed to examine SV2A density in MDD and PTSD as a correlate of synaptic density, and to determine whether ketamine administration will reverse the synaptic loss in vivo in human subjects. To our knowledge, this is the first human study to examine SV2A in vivo in MDD and PTSD and to use the first known drug (ketamine) that rapidly reverses synaptic loss to determine whether ketamine administration could restore some of the structural changes associated with depression and PTSD.

After a screening process to determine eligibility, all subjects will participate in an MRI, and 2-3 PET scans with the administration of ketamine for one of the scans. Cognitive testing and a stress test may also be done on scan days.

DETAILED DESCRIPTION:
The goal of the study is to determine whether there are alterations in synaptic vesicle glycoprotein 2A (SV2A), a protein expressed ubiquitously in synaptic vesicles, in depression and anxiety and whether ketamine, an N-Methyl-D-aspartate (NMDA) antagonist, normalizes SV2A density at time of its greatest anti-depressant response. This study will conduct an examination of SV2A and associated consequences using neuroreceptor imaging and behavioral techniques for the following aims.

Aim 1: To compare SV2A availability in individuals with MDD, healthy control individuals, bipolar individuals, and individuals with PTSD using APP311 or SDM-8 (aka SynVesT-1) and PET.

Hypothesis 1: This study hypothesizes lower SV2A density in MDD, BD, and PTSD in the prefrontal cortex.

Aim 2: To determine whether ketamine administration alters SV2A density in HC, MDD, and PTSD individuals.

Hypothesis 2: This study hypothesizes administration of ketamine will lead to a significant increase in SV2A density in all subject groups (HC, MDD, and PTSD), and this increase will correlate with antidepressant response in individuals with MDD.

Aim 3: To determine the extent of SV2A density changes after prolonged treatment with ketamine in individuals with depression (n=10).

Hypothesis 3: We hypothesize ketamine treatment will increase SV2A density in these individuals. These are individuals who are undergoing ketamine treatment at Yale, CMHC, or surrounding clinics.

Aim 4: To examine changes in SV2A associated with gender within each psychiatric group.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  1. Subjects will be 18-70 years old,
  2. English speaking,
  3. No other DSM-5 diagnosis present, besides required as below.

Inclusion criteria for depressed subjects:

1. Meet DSM-5 diagnostic criteria for Major Depressive Disorder, and for a current depressive episode.
2. Treatment or non-treatment seeking who understand that this study is for research purposes only.

Inclusion criteria for healthy controls:

1. No current, or history of any DSM-5 diagnosis.

Inclusion criteria for PTSD subjects:

1. Current Post Traumatic Stress Disorder.

Inclusion criteria for bipolar subjects:

1. Meet DSM-5 diagnostic criteria for bipolar disorder.

Inclusion criteria for subjects undergoing ketamine treatment

1. Meet DSM-5 diagnostic criteria for Major Depressive Disorder, and for a current depressive episode, as assessed by structured interview for DSM-5 diagnosis (SCID).
2. Undergoing ketamine treatment.

Exclusion Criteria:

1. History of significant medical illness that would contraindicate study participation based on above criteria and PI/MD history review.
2. Lifetime history of neurologic abnormality including seizure disorder, cerebrovascular or neoplastic lesion, neurodegenerative disorder, or significant head trauma resulting in post-traumatic amnesia >24 hours.
3. Full scale IQ lower than 70.
4. Contraindication to MRI scanning including claustrophobia and presence of a ferromagnetic object, including orthodontic braces. All participants will be screened for metal objects by the same methods used for routine clinical MRI scanning.
5. Pregnancy or breast-feeding.
6. Met DSM-5 criteria for mild substance use disorder (except nicotine and marijuana) within the past 6 months or met DSM-5 criteria for moderate to severe substance use disorder within the past year.
7. Claustrophobia.
8. Current psychosis, active suicidal or homicidal ideation.
9. Positive urine toxicology screen (except for marijuana).
10. Contraindications to PET (e.g., past or current diagnosis of cancer, poor venous access for placement of venous lines).
11. History of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure.
12. Previous or anticipated radiation exposure at work within one year of the proposed research PET scans that precludes study participation.
13. Blood pressure >130/80 (for Aim 2, ketamine challenge); blood pressure >140/90 (non-ketamine groups).
14. Arterial line exclusion: History of a bleeding disorder or currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto).
15. Arterial line exclusion: Blood donation within eight weeks of the start of the study.
16. Current diagnosis of MDD or PTSD with psychotic features.
17. Hematocrit levels below 35 mg/dl, and/or hemoglobin levels below 10 mg/dl.
18. Weight under 110 lbs for subjects who will participate in portions of this study for which the blood draw is at or above a typical blood donation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2016-04; Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evidence of synaptic changes in psychiatric disorders confirmed by PET data. | Through study completion date, an average of 5 years.
Evidence of synaptic density at time of its greatest anti-depressant response in psychiatric disorders confirmed with PET data. | Through study completion date, an average of 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Esterlis, PhD, Principal Investigator — Yale University
Locations (1):
- PET Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No